CLINICAL TRIAL: NCT05117138
Title: Safety and Efficacy of Chimeric Antigen Receptor T Lymphocytes for Patients With Intermediate and Advanced Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHSW016
Record Dates: First submitted 2021-09-06; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSCLC/HNSCC：AMT-116 CAR-T cells (Experimental): Patients with moderate or far advanced non-small cell lung carcinomav or head and neck Squamous Cell Carcinoma.
  Interventions: Biological: AMT-116 CAR-T cells
- MEL：AMT-253 CAR-T cells (Experimental): Patients with moderate or far advanced melanoma.
  Interventions: Biological: AMT-253 CAR-T cells

INTERVENTIONS:
Biological: AMT-116 CAR-T cells — 1. Classical "3+3" dose escalation will be applied to 9 subjects with moderate or far advanced non-small cell lung carcinoma (NSCLC) enrolled.
  2. Classical "3+3" dose escalation will be applied to 9 subjects with moderate or far advanced head and neck Squamous Cell Carcinoma (HNSCC) enrolled.
  Arms: NSCLC/HNSCC：AMT-116 CAR-T cells
Biological: AMT-253 CAR-T cells — 1.The classic "3 + 3" dose escalation will be applied to 9 selected subjects with moderate or far advanced melanoma by intravenous drip.
  2.3 ~ 6 patients with intermediate and advanced melanoma will be injected intratumorally at a dose of ≤ 1 × 10^8 cells.
  3.3 ~ 6 patients with operable advanced melanoma will be treated with postoperative adjuvant treatment at a dose of ≤ 1 × 10^8 cells ≤ intravenous drip on Day 1 of each 42 days cycle (8 cycle maximum).
  Arms: MEL：AMT-253 CAR-T cells

SUMMARY:
This was a single arm, open-label, single center, cohort study to determine the efficacy and safety of AMT-116 CAR-T cells in patients with moderate or far advanced non-small cell lung carcinoma (NSCLC) and squamous cell cancer of the head and neck (HNSCC)，AMT-253 CAR-T cells in patients with moderate or far advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, both men and women, and the survival period is more than 6 months.
* At least one assessable focus, failure of previous multi-line treatment or stable condition after treatment.
* Patients with melanoma confirmed by histopathology, patients with non-small cell lung cancer(squamous carcinoma) and head and neck squamous cell carcinoma.
* The surgically removed pathological tissue can be used for immunohistochemical detection of target protein (paraffin section should be within 5 years), and the positive expression of target protein in line with pathological diagnosis (immunohistochemical staining + + or + + +).
* Sufficient venous access for blood sampling and venous blood sampling, no contraindications for lymphocyte collection.
* Routine blood examination: white blood cell count (WBC) ≥ 3 × 10^9 / L, lymphocyte count (ly) ≥ 0.8 × 10^9 / L, hemoglobin (HB) ≥ 90g / L, platelet (PLT) ≥ 80 × 10^9/L.
* Liver and kidney function: alanine aminotransferase and aspartate aminotransferase < 3 ULN, total bilirubin (TBIL) < 1.5 ULN, serum creatinine (SCR) < 2 ULN.
* The subjects voluntarily joined the study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Active hepatitis B or hepatitis C virus, HIV infection, or other unhealed active infections.
* Patients with second tumor.
* Patients previously treated with car-t cells.
* Requiring long-term use of immunosuppressants for any reason.
* Any serious and uncontrolled systemic autoimmune disease or any unstable systemic disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease and temporal arteritis.
* Subjects with severe heart, lung, liver and kidney dysfunction or severe lung diseases.
* Current systemic use of steroid cells (except for recent or current use of inhaled steroids).
* Pregnant and lactating subjects.
* Allergic to immunotherapy and related cells.
* Subjects with a history of organ transplantation or waiting for organ transplantation.
* After evaluation, the investigator considered that the subjects were unable or unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 weeks
Overall Response Rate (ORR) | 24 weeks
One year recurrence rate | 24 weeks

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | 24 weeks
Relapse Free Survival(RFS) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No